CLINICAL TRIAL: NCT05473377
Title: Developing a Computerized Testing System for Measuring Motor and Sensory Integrative Functions in School-aged Children With Intellectual Disabilities
Brief Title: Computerized Testing System for Measuring Motor and Sensory Integrative Functions in Intellectual Disabilities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-SV(I)-20210116
Record Dates: First submitted 2022-07-05; First posted 2022-07-25 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the motor and sensory integrative functions (MSI) is a key component of an overall health and functional evaluation for school-aged children with intellectual disabilities (ID). An efficient and in-depth understanding of the students' motor and sensory integrative functions can help the school teachers implementing appropriate curriculum, monitoring the progress, managing the classroom, and further enhancing the overall learning for school-aged students with ID.

Therefore, in this 2-year project, the investigators will develop a mobile application (APP) testing system for assessing Motor and Sensory Integrative Functions in School-aged Children with Intellectual Disabilities (MSI-ID) to overcome the aforementioned challenges.

The investigators will determine whether the MSI-ID is efficient and psychometrically robust. Around150 to 200 school-aged children with ID will be recruited for this study.

DETAILED DESCRIPTION:
Background and purposes: Assessment of the motor and sensory integrative functions (MSI) is a key component of an overall health and functional evaluation for school-aged children with intellectual disabilities (ID). The ability of students with ID to perform age-appropriate motor tasks and adaptive behaviors (end product of sensory integration) can help determine the long-term effects of special education curriculum/interventions and the quality of an overall school-based rehabilitation program.

However, several challenges exist in measuring MSI for school-aged children with ID. First, most measures of MSI vary in content (domains), causing difficulty in the selection of relevant MSI measures. Second, most measures of MSI lack robust evidence of psychometric properties (e.g., reliability and responsiveness). Third, the minimal important difference (MID) and minimal detectable change (MDC) of most MSI measures for ID are largely unknown, which limits the interpretation of change scores in schools and clinical settings. Fourth, most MSI measures are time-consuming to administer, placing a burden of administration on both teachers/therapists and children. Finally, all the measures were developed in western countries and their use has not yet been validated for ID populations in Taiwan. An efficient and in-depth understanding of the students' motor and sensory integrative functions can help the school teachers implementing appropriate curriculum, monitoring the progress, managing the classroom, and further enhancing the overall learning for school-aged students with ID. A validated and convenient computerized testing system is urgently needed.

The Rasch model is useful in developing precise measures. Furthermore, a computerized adaptive testing (CAT) system can provide efficient measurements. Therefore, in this 3-year project, the investigators will develop a mobile APP testing system for assessing Motor and Sensory Integrative Functions in School-aged Children with Intellectual Disabilities (MSI-ID) to overcome the aforementioned challenges. The investigators will determine whether the MSI-ID is efficient and psychometrically robust. In our previous research (109WFD2110353), the investigators have established the item banks for 3 core domains of MSI (i.e., gross motor, fine motor, and sensory integration) and completed administering on 100 school-aged children with various levels of ID severity and age.

Method: In the first year, the investigators will examine the model fitting of the established items and calibrate the item characteristics with Rasch modeling. Then, the MSI-ID (a tablet personal computer version) will be developed. The investigators will perform a simulation study to determine the performance (e.g., efficiency) of the MSI-ID. In the second year, the investigators will validate the MSI-ID. The tablet MSI-ID will be administered on 150 school-aged children with ID to validate its efficiency (i.e., feasibility and administration time) and psychometric properties (including reliability, validity, responsiveness, and minimal detectable change). A MSI-ID APP will be developed to facilitate the accessibility and utility and the testing system.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 and 15 years
* a diagnosis of ID determined by the board-certified physicians at local designated hospitals according to the standards put forth by the International Classification of Diseases, 10th revision, clinical modification (ICD-10 codes)
* absence of serious emotional , behavioral disturbances or any other major disease affecting premorbid sensory processing and motor functions (e.g., cardiovascular diseases. muscular dystrophy, etc.)
* participation in occupational therapy program at the time of research.

Exclusion Criteria:

-Severe emotional disturbances.

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: To ensure selection of children with major diagnoses of ID and age range in this study, a stratified sampling method will be used to recruit children for psychometric studies. Two stratifying variables will be considered. One is the severity of ID identified in ICD-10 (2 levels: borderline/mild, and moderate/severe). The other is the age band (5 strata: 6:0-6:11, 7:0-7:11, 8:0-10:11, 10:0-11:11, and 12:0-14:11 years).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency- Second Edition | pretest: within the first month of the study
  The Bruininks-Oseretsky Test of Motor Proficiency- Second Edition assesses proficiency in four motor-area composites: fine manual control composite, manual coordination composite, body coordination composite, and strength and agility composite. The four composite scores are combined to yield a total motor composite score. The average age-adjusted scale scores for subtests are 15 (S.D. = 5), whereas composites are derived by summing the subtest scale scores and converting them to a quotient with a mean of 100 and a S.D. of 15. The minimum is 20, and the maximum is 80. Higher score means better outcome
Bruininks-Oseretsky Test of Motor Proficiency- Second Edition | posttest：6 months after the pretest
  The Bruininks-Oseretsky Test of Motor Proficiency- Second Edition assesses proficiency in four motor-area composites: fine manual control composite, manual coordination composite, body coordination composite, and strength and agility composite. The four composite scores are combined to yield a total motor composite score. The average age-adjusted scale scores for subtests are 15 (S.D. = 5), whereas composites are derived by summing the subtest scale scores and converting them to a quotient with a mean of 100 and a S.D. of 15. The minimum is 20, and the maximum is 80. Higher score means better outcome
Sensory Profile | pretest: within the first month of the study
  The Sensory Profile is a parent report measure of behaviors associated with abnormal responses to sensory stimuli for children 5-10 years of age. The Sensory Profile consists of 125 items grouped into three main sections: Sensory Processing, Modulation, and Behavioral and Emotional Responses. Items are scored from always (1) to never (5). The minimum is 125, and the maximum is 575. Higher scores indicate worse outcome. Scores at or above the mean are considered ''typical''; scores of 1 standard deviation below the mean for the typical reference sample are reported as a ''probable difference'', and scores at 2 standard deviations below the mean for the typical reference sample are reported as a ''definite difference''. Internal consistency of sections ranged from 0.47 to 0.90, and the standard error of measurement ranged from 1.13 to 2.81.90 The moderate correlations between the Sensory Profile and the School Function Assessment also supported its validity.
Sensory Profile | posttest: 6 months after the pretest
  The Sensory Profile is a parent report measure of behaviors associated with abnormal responses to sensory stimuli for children 5-10 years of age. The Sensory Profile consists of 125 items grouped into three main sections: Sensory Processing, Modulation, and Behavioral and Emotional Responses. Items are scored from always (1) to never (5). The minimum is 125, and the maximum is 575. Higher scores indicate worse outcome. Scores at or above the mean are considered ''typical''; scores of 1 standard deviation below the mean for the typical reference sample are reported as a ''probable difference'', and scores at 2 standard deviations below the mean for the typical reference sample are reported as a ''definite difference''. Internal consistency of sections ranged from 0.47 to 0.90, and the SEM ranged from 1.13 to 2.81.90 The moderate correlations between the Sensory Profile and the School Function Assessment also supported its validity.
Test of Visual Perceptual Skills, Third Edition | pretest: within the first month of the study
  The Test of Visual Perceptual Skills assesses visual perception for individuals aged 4-18 years 11 months in seven comprehensive subtests: visual discrimination, visual memory, visual spatial relationship, visual form constancy, visual sequential memory, visual figure-ground, and visual closure. The minimum is 55 and the maximum is 145, higher score means better outcome.
Test of Visual Perceptual Skills, Third Edition | posttest：6 months after the pretest
  The Test of Visual Perceptual Skills assesses visual perception for individuals aged 4-18 years 11 months in seven comprehensive subtests: visual discrimination, visual memory, visual spatial relationship, visual form constancy, visual sequential memory, visual figure-ground, and visual closure. The minimum is 55 and the maximum is 145, higher score means better outcome.
Cognitive/Behavioral Tasks Performance Scale (CBTPS) of School Function Assessment | pretest: within the first month of the study
  The School Function Assessment is a judgment-based assessment that measures a student's performance of functional tasks that support his or her participation in both academic and social school-related activities for students in grades kindergarten to 6th grade. The Cognitive/Behavioral Tasks Performance Scale (CBTPS) was used as an external criterion for clinically relevant change in the present study. The CBTPS include 121 items under 9 domains: functional communication, memory and understanding, following social conventions, compliance with adult directives and social rules, task/behavior completion, positive interaction, behavior regulation, personal care awareness, and safety. The activities are rated on a scale of 1 to 4, where 1 = does not perform, 2 = partial performance, 3 = inconsistent performance, and 4 = consistent performance. The minimum is 121, and the maximum is 484. Higher scores mean better outcome.
Cognitive/Behavioral Tasks Performance Scale (CBTPS) of School Function Assessment | posttest: 6 months after the pretest
  The School Function Assessment is a judgment-based assessment that measures a student's performance of functional tasks that support his or her participation in both academic and social school-related activities for students in grades kindergarten to 6th grade. The Cognitive/Behavioral Tasks Performance Scale (CBTPS) was used as an external criterion for clinically relevant change in the present study. The CBTPS include 121 items under 9 domains: functional communication, memory and understanding, following social conventions, compliance with adult directives and social rules, task/behavior completion, positive interaction, behavior regulation, personal care awareness, and safety. The activities are rated on a scale of 1 to 4, where 1 = does not perform, 2 = partial performance, 3 = inconsistent performance, and 4 = consistent performance. The minimum is 121, and the maximum is 484. Higher scores mean better outcome.
Physical Task Performance Scale (PTPS) of School Function Assessment | pretest: within the first month of the study
  The School Function Assessment is a judgment-based assessment that measures a student's performance of functional tasks that support his or her participation in both academic and social school-related activities for students in grades kindergarten to 6th grade. The Physical Task Performance Scale (PTPS) was used as an external criterion for clinically relevant change in the present study. The PTPS consists of 161 items (activities) divided into 12 domains including travel, maintaining and changing positions, recreational movement, manipulation with movement, using materials, set-up and cleanup, eating and drinking, hygiene, clothing management, up/down stairs, written work, and computer and equipment use. The activities are rated on a scale of 1-4 according to their performance level. The minimum is 161, and the maximum is 644. Higher scores mean better outcome.
Physical Task Performance Scale (PTPS) of School Function Assessment | posttest: 6 months after the pretest
  The School Function Assessment is a judgment-based assessment that measures a student's performance of functional tasks that support his or her participation in both academic and social school-related activities for students in grades kindergarten to 6th grade. The Physical Task Performance Scale (PTPS) was used as an external criterion for clinically relevant change in the present study. The PTPS consists of 161 items (activities) divided into 12 domains including travel, maintaining and changing positions, recreational movement, manipulation with movement, using materials, set-up and cleanup, eating and drinking, hygiene, clothing management, up/down stairs, written work, and computer and equipment use. The activities are rated on a scale of 1-4 according to their performance level. The minimum is 161, and the maximum is 644. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yee-Pay Wuang, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Dept of Occupational Therapy, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Haley SM, Ni P, Ludlow LH, Fragala-Pinkham MA. Measurement precision and efficiency of multidimensional computer adaptive testing of physical functioning using the pediatric evaluation of disability inventory. Arch Phys Med Rehabil. 2006 Sep;87(9):1223-9. doi: 10.1016/j.apmr.2006.05.018. PMID 16935059
- See also: Measurement precision and efficiency of multidimensional computer adaptive testing of physical functioning using the pediatric evaluation of disability inventory. — https://pubmed.ncbi.nlm.nih.gov/16935059/